CLINICAL TRIAL: NCT06350994
Title: Early Assessment of Cardiac Function After Treatment With CAR-T Cells
Acronym: Cardio CAR-T
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230625; IDRCB 2023-A01957-38 (Other: ANSM)
Record Dates: First submitted 2024-02-21; First posted 2024-04-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Car T- Cell; Hematologic Malignancy; Acute Lymphoblastic Leukemia; Lymphoma, B-Cell; Multiple Myeloma
Keywords: CAR-T cells; Hematological malignancies; Cardiomyopathy; Cardiotoxicity; Pharmacovigilance
MeSH Terms: conditions — Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell; Multiple Myeloma; Cardiomyopathies; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cardio CAR-T: Transthoracic bedside echocardiography

SUMMARY:
CAR-T cells (Chimeric Antigen Receptor) are a new immunotherapy, based on the genetic modification of autologous T lymphocytes. CAR-T cell therapy is not devoid of complications.

Among the most frequent complications are the risk of infection, cytokine release syndrome (CRS) and neurotoxicity. Nevertheless, some authors have reported serious acute cardiac events in a limited number of patients, often contemporaneous with CRS or sepsis, questioning the imputability of CAR-T cells in this heart disease.

This study aims to estimate the incidence of a possible early cardiotoxicity associated with CAR-T cells.

The main endpoint will be the change in cardiac function (LVEF: left ventricular ejection fraction) assessed by ultrasound between the pre CAR-T assessment and the early post CAR-T ultrasound (D3-D5).

DETAILED DESCRIPTION:
CAR-T cells (Chimeric Antigen Receptor) represent a new form of immunotherapy, based on the genetic modification of autologous T lymphocytes collected after apheresis, allowing the recognition of a tumor antigen apart from the presentation by the major complex of histocompatibility (MHC). Treatment with CAR-T cells constitutes a major therapeutic advance in patients with refractory hematological malignancies.

Nevertheless, CAR-T cell therapy is often associated with severe complications leading them to the ICU in >25%.

Among the most frequent complications are the risk of infection cytokine release syndrome (CRS)and neurotoxicity. A recent study reported serious acute cardiac events in the days following the administration of CAR-T cells in 6.5% of patients (12/187). In this work, patients did not benefit from systematic early echocardiography, but only in the event of CRS grade ≥2 or symptoms, with a risk of underdiagnosis of asymptomatic forms. Since the vast majority of reported cases are contemporaneous with CRS or sepsis, the imputability of CAR-Ts in this heart disease is debated.

The Cardio CAR-T study aims to investigate a possible early cardiac toxicity of CAR-T cells, screened by transthoracic echocardiography at the patient's bedside, between D3 and D5 after injection of CAR-T cells (period at which the inflammatory complications of this treatment occur in the majority of cases) associated with the description of routine examinations (BNP, Troponin and ECG) and cytokine analyses.

This pilot descriptive study would answer 2 questions:

* What are the incidence and characteristics of acute cardiac toxicity (clinical and subclinical) of CAR-T cells and their association with CRS?
* Is there a link between cardiac toxicity and the intensity of the cytokine inflammatory response? This makes it possible to provide new pathophysiological elements on the existence of a heart disease directly caused by the inflammatory storm, applicable to other areas such as septic shock, ischemia-reperfusion or major surgery.

ELIGIBILITY:
Inclusion Criteria:

* CAR-T cells infusion received within 3 to 5 days before the echocardiography
* Pre-therapeutic cardiac assessment (in accordance with the recommendations and standard care protocol in force in the hematology department of Saint-Antoine Hospital): Echocardiography and EKG before conditioning and infusion of CAR -T cells,
* Not opposed to participating in research.
* Patient affiliated to a social security system or beneficiary of the "state medical insurance help" (namely aide médicale d'état).

Exclusion Criteria:

* Opposition or consent withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years old) receiving CAR-T cell therapy for hematological malignancies (acute lymphoblastic -B cell leukemia, lymphoma and multiple myeloma) hospitalized in hematology department or in intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Estimation of the incidence of possible early CAR-T cells infusion-induced cardiotoxicity | 5 days and 3 months
  Transthoracic bedside echocardiographic evaluation of the LVEF.

SECONDARY OUTCOMES:
Characterization of the putative CAR-T cells infusion-induced cardiotoxicity: incidence, phenotype, clinical, rhythmic and biological manifestations | 5 days and 3 months
  Transthoracic bedside echocardiographic evaluation of the LVEF, EKG, biologicals (troponin, BNP).
Determination of its possible association with a cytokine release syndrome and the levels of inflammatory biomarkers from the analysis of the serum library of these patients | 5 days and 3 months
  Multiplex bioassays for immune-inflammatory biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie JOFFRE, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Critical care medicine department, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided